CLINICAL TRIAL: NCT02155790
Title: A Safety and Performance Study of Renal Denervation by Neurolysis Using the Ablative Solutions Inc. Peregrine System™ Infusion Catheter
Brief Title: The Peregrine Study: A Safety and Performance Study of Renal Denervation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablative Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASI 12-001
Record Dates: First submitted 2014-05-27; First posted 2014-06-04 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hypertension
Keywords: safety, performance, hypertension, renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Denervation by Neurolysis (Experimental): Infusion of 0.3 ml of dehydrated alcohol (96%-98%) into the peri-adventitial space of the renal artery, to achieve renal denervation by Neurolysis, via three simultaneous deployed needles, situated at the distal end of the Peregrine System Infusion Catheter.
  Interventions: Device: The Peregrine System Infusion Catheter

INTERVENTIONS:
Device: The Peregrine System Infusion Catheter — The ASI catheter is inserted bilaterally into the renal arteries and a specified amount of a neurolytic agent is inserted into the vessel walls.
  Other Names: Renal denervation using a neurolytic agent

SUMMARY:
The Ablative Solutions, Inc. Peregrine System Infusion Catheter is a catheter-based device which is intended to be used to ablate the afferent and efferent sympathetic nerves serving the kidneys. The catheter is typically inserted via the femoral artery, steered into the renal artery, and then delivers, by infusion from its distal end, a neurolytic agent. This targets the nerve bundles, which are in the adventitia - a sheath surrounding the artery. The aim is to reduce blood pressure in cases of resistant hypertension - seriously elevated blood pressure which does not respond to drug treatment.

DETAILED DESCRIPTION:
There is strong evidence in the published literature that the renal nerves are important contributors to hypertension, and that their ablation does not have adverse side-effects. The literature provides technical, clinical and scientific evidence supporting the use of perivascular renal denervation for a carefully defined patient group.

An existing device (the Ardian Symplicity catheter) has been shown to be safe and effective for achieving perivascular renal denervation by delivery of radiofrequency energy. Perivascular renal denervation by radio-frequency energy delivery is an effective therapy, associated with very low risks. In other contexts, denervation can also be safely and effectively achieved by neurolytic agents.

The objectives of the study are to evaluate the safety and performance of renal denervation by a chemical neurolytic agent delivered into the advential/ periadventitial area of the renal arteries for the purpose of neurolysis, using the Peregrine System Infusion Catheter, in patients with refractory hypertension.

The ASI Peregrine System Infusion Catheter is similar enough to the Ardian Symplicity catheter to enable the use of published data to establish the validity of the design concept of the Peregrine System and estimate the likely levels of risk from side effects. It can be concluded from the literature that the ASI Peregrine System will achieve percutaneous renal denervation with a low risk of procedural complications (comparable to accepted percutaneous interventional therapies) and without long-term impairment of renal artery or kidney function or other serious adverse events.

Chemical denervation is an appropriate treatment for the specified study population of adults who have resistant hypertension despite taking at least 3 anti-hypertensive drugs of different classes including at least one diuretic. In order for the study to be valid, only one chemical neurolytic agent can be used. The Coordinating Investigator has chosen to use dehydrated alcohol (96 - 98% by volume) for therapeutic neurolysis, therefore all participating sites will use this agent. This clinical investigation is intended to provide clinical data that demonstrates the safety and performance of the ASI Peregrine System Infusion Catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, age 18-75, male or female;
2. Patient has a clinic systolic blood pressure ≥ 160 mm Hg (or ≥ 150 mm Hg in type 2 diabetic patients) based on an average of 3 office/clinic measurements taken manually;
3. Patient has a daytime mean systolic pressure ≥135 mm Hg based on 24 hours ambulatory blood pressure monitoring, with >85% valid readings.
4. Patient with resistant hypertension is receiving and adhering to a stable medication regimen of at least 3 anti-hypertensive medications of different classes (for at least 4 weeks), one of which must be a diuretic. The three (or more) - medication regimen must be maximal in terms of dose and tolerability in the judgement of the investigator, such that the next step in blood pressure management would be the addition of a further medication.
5. Patient has an eGFR ≥ 45 mL/min, based on the CKD-EPI equation;
6. Patient has no implanted ICD, pacemaker or neurostimulator or any metallic implant which is not compatible with magnetic resonance imaging. THis is applicable to sites were MRI is planned. Implanted devices are acceptable at sites where CT will be used
7. Patient has optimal renal artery anatomy (no clear abnormalities) based on Investigator's evaluation of CT-angiogram/ or as alternative MR-angiogram and /or renal angiogram including:

   * Single or two renal arteries, if each has a 5-7 mm diameter, respectively (accessory renal arteries are acceptable if diameter is is ≤ 2 mm, which will not be treated)
   * No aneurysms
   * No excessive tortuosity
   * No previous stenting or balloon angioplasty of the renal arteries
   * No previous renal denervation;
8. Patient has provided written informed consent

Exclusion Criteria:

1. Patient has known or suspected secondary hypertension;
2. Patient has type 1 diabetes mellitus;
3. Patient requires chronic oxygen support;
4. Patient has primary or secondary pulmonary hypertension;
5. Patient has a known bleeding diathesis.
6. Patient has thrombocytopenia (platelet count <100,000 platelets/µL;
7. Patient is pregnant or nursing or planning to become pregant;
8. Patient has significant imaging-assessed renovascular abnormalities including short length main renal artery (< 10mm) and renal artery stenosis >60% of the normal diameter segment;
9. Patient has history of nephrectomy, a single kidney, kidney tumor or urinary tract obstruction (with potential for hydronephrosis);
10. Patient is known to have a unilateral non-functioning kidney or unequal renal size (>2 cm difference in renal length between kidneys);
11. Patient has a renal transplant;
12. Patient has a history of kidney stones;
13. Patient has a history of heterogeneities in the kidney such as cysts or tumors;
14. Patient has a history of pyelonephritis;
15. Patient has a history of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last six months;
16. Patient has hemodynamically significant valvular heart disease;
17. Patient has heart failure (NYHA III or IV) or has an ejection fraction ≤ 30%;
18. Patient has a known allergy to contrast media;
19. Patient has a life expectancy of <12 months;
20. Patient is currently enrolled in other potentially confounding research, i.e., another therapeutic or interventional research trial. Patients enrolled in observational registries may still be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Vessel dissection or perforation | Immediate post procedure
  Vessel dissection or perforation on immediate post-procedural fluoroscopy
Grade 3 or Grade 4 hemorrhage | During or immediately after procedure
  Grade 3 hemorrhage requiring transfusion or Grade 4 hemorrhage
Cerebrovascular accident | Time of procedure
  Cerebrovascular accident at the time of procedure
Myocardial infarction | Time of procedure
  Myocardial infarction at the time of the procedure
Sudden cardiac death | Time of procedure
  Sudden cardiac death at the time of the procedure
Reduction in the systolic blood pressure | 6 months
  The primary performance endpoint is a reduction in the clinic systolicand diastolic blood pressure following treatment compared to baseline, assessed at 6 months.

SECONDARY OUTCOMES:
Change in eGFR (reduction >25%) | baseline to 6 months
  Proportion of patients with a decline in eGFR by >25% from baseline to 6 months follow-up
New renal arterial stenosis >60% | 6 months
  New renal arterial stenosis >60% from baseline confirmed by the same method used at baseline
Mean change in serum creatinine | post baseline visits at 7d,1 mo,3mo,6mo,12mo,24mo
  Change in serum creatinine
Adverse events | post baseline visits at 7d,1 mo,3mo,6mo,12mo,24moprocedure and each of the follow-up time periods
  Adverse events - device and non-device related
Changes in antihypertensive medications | post baseline visits at 7d,1 mo,3mo,6mo,12mo,24moeach of the follow-up visits
  The addition of new antihypertensive drugs will be considered an intensification of the antihypertensive regimen.
  Discontinuation of one or more of the baseline antihypertensive medications without an increase in dose of remaining drugs or addition of new drugs will be considered a reduction in antihypertensive drug regimen.
Changes in ambulatory blood pressure measurements | post baseline visits at 7d,1 mo,3mo,6mo,12mo,24mo
  Ambulatory blood pressures will be reported to determine if they follow a similar patter to the clinic blood pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Wojakowski, Prof.MD.PhD, Principal Investigator — American Hospitals Poland
Locations (3):
- Na Homolce Hospital, Prague, Czechia
- Poland (2):
  - American Heart of Poland, Tychy
  - American Heart of Poland, Ustroń